CLINICAL TRIAL: NCT02132689
Title: Comparison of Thrombgolytic and Anticoagulation Therapy in Submassive Pulmonary Embolism in Context of Pulmonary Hypertension, Right Heart Failure and Patient Functional Ability
Brief Title: Comparison of Thrombgolytic and Anticoagulation Therapy in Submassive Pulmonary Embolism
Acronym: CONTACT-SPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Municipal Hospital Ostrava Fifejdy (Unknown); Silesian Hospital Opava (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-KVO-3
Record Dates: First submitted 2014-04-28; First posted 2014-05-07 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Embolism
Keywords: Moderate Risk Acute Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator; Thrombolytic Therapy; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Actilyse (Active Comparator): Thrombolytic therapy: Patients treated with initial thrombolytic therapy (Actilyse) followed with anticoagulant therapy (unfractionated/low-molecular weight heparin).
  Interventions: Drug: Actilyse (Thrombolytic therapy); Drug: Heparine (Standard anticoagulation therapy)
- UHF/LMWH (Active Comparator): Anticoagulation therapy: Patients treated with anticoagulation therapy only (unfractionated/low-molecular weight heparin).
  Interventions: Drug: Heparine (Standard anticoagulation therapy)

INTERVENTIONS:
Drug: Actilyse (Thrombolytic therapy)
  Other Names: Actilyse
  Arms: Actilyse
Drug: Heparine (Standard anticoagulation therapy)
  Other Names: unfractionated/low-molecular weight heparine

SUMMARY:
Currently there is no clear guidance for the treatment of moderate risk of pulmonary embolism. The aim of the study is to compare two different therapeutic modalities - standard anticoagulation versus thrombolytic treatment followed by anticoagulation in standard regimen as stated in the pulmonary embolism guidelines.

DETAILED DESCRIPTION:
Standard treatment of moderate risk pulmonary embolism constitutes of sole anticoagulation therapy. In case of troponin positivity and/or echocardiographic findings as i.e. thrombi in RV thrombolytic therapy should be considered. The aim of this trial is to compare the two treatment modalities in their ability to reduce/predict 12 month end-point: pulmonary hypertension, right ventricular failure, exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* moderate risk pulmonary embolism as defined by the European Society of Cardiology /ESC/ guidelines
* signed informed consent

Exclusion Criteria:

* patient not willing to sigh informed consent
* absolute contraindication of thrombolysis
* inability to obtain meaningfull echocardiographic images¨
* pulmonary arterial hypertension
* known right ventricular failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical manifestations of right ventricular failure and pulmonary hypertension and cardiovascular-related death | 12 months
  The primary outcome of the study is to follow clinical manifestations of right ventricular failure (assessed according to the New York Heart Association /NYHA/ classification).
Pulmonary hypertension | 12 months
  The primary outcome of the study is to follow pulmonary hypertension (measured in mmHg).
Cardiovascular-related deaths | 12 months
  The primary outcome of the study is to follow the number of cardiovascular-related deaths within the time frame of 12 months.

SECONDARY OUTCOMES:
Echocardiographic manifestations of right ventricular failure and pulmonary hypertension. | 12 months
  The secondary outcome measure of the study is to follow echocardiographic manifestations of right ventricular failure (TdiSm).

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Stancik, MD, Principal Investigator — Department of Cardiology, University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Silesian Hospital Opava, Opava
  - University Hospital Ostrava, Ostrava-Poruba